CLINICAL TRIAL: NCT02138552
Title: Phase II Study to Assess Bacterial Count Reduction of Three Octenidine Mouthwash Concentrations in Comparison to a Placebo in Patients With Mild Gingivitis
Brief Title: Dose Finding Study to Assess Octenidine Mouthwash Concentrations in Comparison to Placebo
Acronym: OML0113
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Schülke & Mayr GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-002708-14
Record Dates: First submitted 2013-11-11; First posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — octenidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- OCT 0.1% vs. Placebo (Active Comparator): 0.1 % Octenidine dihydrochloride vs. Placebo (0.9 % sodium chloride solution)
  Interventions: Drug: Octenidine dihydrochloride; Drug: Placebo
- OCT 0.15% vs. Placebo (Active Comparator): 0.15 % Octenidine dihydrochloride vs. Placebo (0.9 % sodium chloride solution)
  Interventions: Drug: Octenidine dihydrochloride; Drug: Placebo
- OCT 2.0% vs. Placebo (Active Comparator): 0.2 % Octenidine dihydrochloride vs. Placebo (0.9 % sodium chloride solution)
  Interventions: Drug: Octenidine dihydrochloride; Drug: Placebo

INTERVENTIONS:
Drug: Octenidine dihydrochloride — Mouthrinsing - comparison of different dosages of Octenidine dihydrochloride over 4 days vs. Placebo
Drug: Placebo — Mouthrinsing - comparison of different dosages of Octenidine dihydrochloride over 4 days vs. Placebo

SUMMARY:
The objective of this clinical trial is to identify the most efficacious octenidine dihydrochloride concentration regarding bacterial count reduction in comparison to a placebo in the oral cavity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild gingivitis (mean GI: 0.2 - 1.0)
* Patients with complete natural "Ramfjord-teeth" or their replacement teeth
* Caucasian
* Signed Informed Consent

Exclusion Criteria:

* Patients with severe systemic diseases (diabetes, hepatitis, HIV, tuberculosis, cancer)
* Patients who require endocarditis prophylaxis for dental examination and treatment
* Caries requiring treatment (e.g. caries with cavity) or other oral diseases (incl. gingival hyperplasia, diseases of the oral mucosa, periodontal screening index PSI > 2)
* Patients with orthodontic appliances and removable dentures
* Patients treated with antibiotics less than 3 months prior to the baseline examination at V1 and/or such a treatment planned for the duration of the trial
* Patients chronically treated with steroids
* Patients who suffer from xerostomia
* Patients who regularly smoke more than 10 cigarettes per day
* Patients who have a known hypersensitivity or allergy to the test product and its ingredients or to medications that have a similar chemical structure
* Participation of the patient in another clinical trial within the last four weeks before enrollment in this trial
* Incapability of assessing essence and possible consequences of the trial (e.g. alcoholism)
* Pregnant or breastfeeding women
* Women with childbearing potential except those who fulfill the following criteria:

  * Post-menopausal (12 month of natural amenorrhoea or 6 months of amenorrhoea with Serum FSH > 40 U/ml)
  * Postoperative (6 weeks after bilateral ovariectomy with or without hysterectomy)
  * Continuous and correct application of a contraception method with a Pearl Index < 1% (e.g. implants, depots, oral contraceptives, intrauterine device - IUD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Bacterial count reduction in saliva after a single application of OML in comparison to placebo application | After 1 minute of rinsing
  Bacterial count reduction is measured at V1 (Verum/Placebo) and V3 (Placebo/Verum) in a blinded cross-over design

SECONDARY OUTCOMES:
Mean plaque index (PI) | After 5 days of application
  PI is measured at V2 (Verum/Placebo) and V4 (Placebo/Verum) in a blinded cross-over design
Change in mean gingival index (GI) | After 5 days of application
  GI is measured at V1/V2 (Verum/Placebo) and V3/V4 (Placebo/Verum) in a blinded cross-over design
Evaluation of taste and flavour (questionnaire) | After 5 days of application
AEs and SAEs | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Lorenz, Dr., Study Director — Poliklinik für Parodontologie Med. Fakultät C. G. Carus der TU Dresden
Locations (2):
- Germany (2):
  - Poliklinik für Parodontologie Med. Fakultät C. G. Carus der TU Dresden, Dresden
  - Abteilung für Parodontologie in der Poliklinik für Zahnerhaltung und Parodontologie der Universität Würzburg, Würzburg